CLINICAL TRIAL: NCT00404547
Title: An Open-Label Randomized, Multicenter Study in Patients With Asthma to Evaluate the Effectiveness of Alvesco® (Ciclesonide) Compared to Asthma Usual Care in a Primary Practice Setting
Brief Title: Asthma Care With Alvesco® (Ciclesonide) in Primary Care in Adults - The ACCEPT-study (BY9010/CA-102)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY9010/CA-102
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Alvesco®; Ciclesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alvesco (Active Comparator): Alvesco 320mcg / Alvesco 640mcg
  Interventions: Drug: Ciclesonide
- Usual Care (Active Comparator)
  Interventions: Drug: Usual Care Inhaled Glucocorticosteroids

INTERVENTIONS:
Drug: Ciclesonide — Asthma Care with Alvesco
  Arms: Alvesco
Drug: Usual Care Inhaled Glucocorticosteroids — Usual asthma care and dosage as chosen by the Primary Care Physician including inhaled steroid treatment
  Arms: Usual Care

SUMMARY:
The purpose of this study is to investigate the effectiveness of Alvesco® (Ciclesonide) compared with usual asthma care in the primary care setting. Patients with a history of asthma for at least 6 months and who, in the opinion of the physician, meet the clinical requirements for treatment with inhaled steroids (ICS) will be enrolled. They will either receive Alvesco® or usual care.

ELIGIBILITY:
Main inclusion criteria:

* Written informed consent
* 18 years or older with diagnosis of asthma for at least 6 months
* Clinically stable asthma at the time of study enrollment
* Clinical requirements for treatment with ICS as outlined in the Canadian Asthma Consensus Guidelines
* If patients are currently on ICS, the dose must be stable for 3 months and they must be willing to switch

Main exclusion criteria:

* On combination therapy (ICS + long acting beta-2-agonist) for asthma in the past 3 months or require combination therapy
* Severe asthma, one or more asthma exacerbations in the last 3 months requiring hospitalization or emergency room visit, or patients who have used systemic steroids more than 3 times in the past 6 months or who are currently using systemic steroids
* Mild asthma requiring short acting beta-2-agonists only
* Patients with a contraindication to ICS therapy
* Any other disease or medical condition requiring further clinical evaluation, which in the opinion of the Primary Care Practitioner may interfere with the clinical study or interfere with the diagnosis of asthma.
* Pregnancy, breast feeding, intention to become pregnant during the course of the study or lack of safe contraception in pre-menopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1121 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (99):
- Canada (99):
  - "Altana Pharma/Nycomed", Abbotsford
  - "Altana Pharma/Nycomed", Ajax
  - "Altana Pharma/Nycomed", Alma
  - "Altana Pharma/Nycomed", Anjou
  - "Altana Pharma/Nycomed", Barrie
  - "Altana Pharma/Nycomed", Brampton
  - "Altana Pharma/Nycomed", Brossard
  - "Altana Pharma/Nycomed", Burnaby
  - "Altana Pharma/Nycomed", Cacouna
  - "Altana Pharma/Nycomed", Calgary
  - "Altana Pharma/Nycomed", Cambridge
  - "Altana Pharma/Nycomed", Collingwood
  - "Altana Pharma/Nycomed", Conception Bay S
  - "Altana Pharma/Nycomed", Cornwall
  - "Altana Pharma/Nycomed", Corunna
  - "Altana Pharma/Nycomed", Courcelette
  - "Altana Pharma/Nycomed", Delta
  - "Altana Pharma/Nycomed", Dolbeau-Mistassini
  - "Altana Pharma/Nycomed", Edmonton
  - "Altana Pharma/Nycomed", Etobicoke
  - "Altana Pharma/Nycomed", Fort Erie
  - "Altana Pharma/Nycomed", Gatineau
  - "Altana Pharma/Nycomed", Gatineau (Sector Hull)
  - "Altana Pharma/Nycomed", Grand Falls
  - "Altana Pharma/Nycomed", Greater Sudbury
  - "Altana Pharma/Nycomed", Halifax
  - "Altana Pharma/Nycomed", Harrow
  - "Altana Pharma/Nycomed", Hastings
  - "Altana Pharma/Nycomed", Hull
  - "Altana Pharma/Nycomed", Joliette
  - "Altana Pharma/Nycomed", Jonquière
  - "Altana Pharma/Nycomed", Kamloops
  - "Altana Pharma/Nycomed", Kentville
  - "Altana Pharma/Nycomed", Keswick
  - "Altana Pharma/Nycomed", Kingston
  - "Altana Pharma/Nycomed", Kirkland
  - "Altana Pharma/Nycomed", LaSalle
  - "Altana Pharma/Nycomed", Laval
  - "Altana Pharma/Nycomed", London
  - "Altana Pharma/Nycomed", Milton
  - "Altana Pharma/Nycomed", Mississauga
  - "Altana Pharma/Nycomed", Moncton
  - "Altana Pharma/Nycomed", Montreal
  - "Altana Pharma/Nycomed", Mount Pearl
  - "Altana Pharma/Nycomed", Niagara Falls
  - "Altana Pharma/Nycomed", North Bay
  - "Altana Pharma/Nycomed", North Sydney
  - "Altana Pharma/Nycomed", North Vancouver
  - "Altana Pharma/Nycomed", North York
  - "Altana Pharma/Nycomed", Oakville
  - "Altana Pharma/Nycomed", Oshawa
  - "Altana Pharma/Nycomed", Ottawa
  - "Altana Pharma/Nycomed", Penticton
  - "Altana Pharma/Nycomed", Perth-Andover
  - "Altana Pharma/Nycomed", Point Edward
  - "Altana Pharma/Nycomed", Pointe-Claire
  - "Altana Pharma/Nycomed", Princeville
  - "Altana Pharma/Nycomed", Québec
  - "Altana Pharma/Nycomed", Red Deer
  - "Altana Pharma/Nycomed", Regina
  - "Altana Pharma/Nycomed", Repentigny
  - "Altana Pharma/Nycomed", Richmond
  - "Altana Pharma/Nycomed", Richmond Hill
  - "Altana Pharma/Nycomed", Rimouski
  - "Altana Pharma/Nycomed", Roxton Pond
  - "Altana Pharma/Nycomed", Saint John
  - "Altana Pharma/Nycomed", Saint Romuald
  - "Altana Pharma/Nycomed", Saint-Jérôme
  - "Altana Pharma/Nycomed", Saint-Léonard
  - "Altana Pharma/Nycomed", Saint-Pie
  - "Altana Pharma/Nycomed", Sainte-Catherine
  - "Altana Pharma/Nycomed", Sarnia
  - "Altana Pharma/Nycomed", Saskatoon
  - "Altana Pharma/Nycomed", Scarborough
  - "Altana Pharma/Nycomed", Sherbrooke
  - "Altana Pharma/Nycomed", Shubenacadie
  - "Altana Pharma/Nycomed", St-Bruno
  - "Altana Pharma/Nycomed", St-Jean-sur-Richel
  - "Altana Pharma/Nycomed", St. Catharines
  - "Altana Pharma/Nycomed", St. John's
  - "Altana Pharma/Nycomed", Ste Anne de Bellev
  - "Altana Pharma/Nycomed", Stirling
  - "Altana Pharma/Nycomed", Stouffville
  - "Altana Pharma/Nycomed", Surrey
  - "Altana Pharma/Nycomed", Sydney Mines
  - "Altana Pharma/Nycomed", Thetford-Mines
  - "Altana Pharma/Nycomed", Thornhill
  - "Altana Pharma/Nycomed", Thunder Bay
  - "Altana Pharma/Nycomed", Toronto
  - "Altana Pharma/Nycomed", Vancouver
  - "Altana Pharma/Nycomed", Verdun
  - "Altana Pharma/Nycomed", Victoria
  - "Altana Pharma/Nycomed", West Vancouver
  - "Altana Pharma/Nycomed", Westmount
  - "Altana Pharma/Nycomed", Whitby
  - "Altana Pharma/Nycomed", Windsor
  - "Altana Pharma/Nycomed", Winnipeg
  - "Altana Pharma/Nycomed", Woodstock
  - "Altana Pharma/Nycomed", York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of subjects STARTED is related to the number of randomized subjects (= subjects who were eligible for treatment period). It differs from the number of subjects of the Intention to Treat (ITT) population in Baseline Characteristics and Outcome Measures. The statistical analyses of the Outcome Measures is based on the ITT population.
Groups:
- Alvesco: 320 mcg/day or 640 mcg/day
- Usual Asthma Care and Dosage: as chosen by the Primary Care Physician
Period: Overall Study
Arm/Group | Alvesco | Usual Asthma Care and Dosage
Started | 762 | 359
Completed | 672 | 334
Not Completed | 90 | 25
Not completed — Adverse Event | 39 | 6
Not completed — Withdrawal by Subject | 19 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 20 | 9
Not completed — Lack of compliance | 5 | 1
Not completed — Other | 4 | 0
Not completed — Reason not stated | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvesco | Usual Asthma Care and Dosage | Total
Number analyzed (Participants) | 712 | 345 | 1057
Age, Customized [Mean (Standard Deviation); unit: years] — Basis is the Intention to Treat Population (ITT).
  years | 47.3 (16.3) | 47.2 (16.7) | 47.26 (16.43)
Gender [Count of Participants; unit: Participants] — Basis is the Intention to Treat Population (ITT).
  Participants
    Female | 431 | 232 | 663
    Male | 281 | 113 | 394
Smoking Status [Number; unit: participants] — Basis is the Intention to Treat Population (ITT).
  participants
    Never | 359 | 149 | 508
    Current | 156 | 81 | 237
    Former | 197 | 115 | 312
Duration of Asthma [Mean (Standard Deviation); unit: years] — Basis is the Intention to Treat Population (ITT).
  years | 12.4 (11.3) | 12.8 (11.9) | 12.5 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean of Total Score of Asthma Control Questionnaire (ACQ)
Description: The score of the change from baseline ranges from -6 (=best possible outcome) to 6 (=worst possible outcome).
Time Frame: At the middle and end of the 12 week treatment period
Population: Basis is the ITT population
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Alvesco | Usual Asthma Care and Dosage
Number analyzed (Participants) | 712 | 345
points on a scale | -0.76 (0.97) | -0.37 (0.98)
Statistical Analysis 1: Comparison: Alvesco vs Usual Asthma Care and Dosage; This is an analysis of the change in Asthma Control Questionnaire (ACQ) after 12 weeks of treatment; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Change in Patient Assessment of Asthma Control
Description: Patient assessment of asthma control was assessed at baseline and at week 12 using the question "How would you rate the control of your asthma symptoms?". The change in this assessment was categorized in "Improvement" and "Non-Improvement".
Time Frame: At baseline and at week 12
Population: Basis is the ITT population
Measure: Number; unit: participants
Arm/Group | Alvesco | Usual Asthma Care and Dosage
Number analyzed (Participants) | 712 | 345
participants
  Improvement | 422 | 132
  Non-Improvement | 284 | 209
  Not reported | 6 | 4

3. Secondary Outcome: Assessment of Patient Compliance During the Study
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of Patient Treatment Satisfaction
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The numbers of subjects at risk are based on the Safety Population. It was based on all randomized patients receiving at least one dose of the double-blind study medication after randomization.
Arm/Group | Alvesco | Usual Asthma Care and Dosage
Serious Adverse Events (participants affected / at risk) | 6/741 | 1/346
Other Adverse Events (participants affected / at risk) | 0/741 | 0/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvesco (N=741) | Usual Asthma Care and Dosage (N=346)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days